CLINICAL TRIAL: NCT01433913
Title: Phase II Study of Metformin in a Pre-prostatectomy Prostate Cancer Cohort
Brief Title: Metformin Hydrochloride in Treating Patients With Prostate Cancer Undergoing Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-00243; NCI-2012-00243 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000712087; UARIZ-UAZ10-16-01; 11-0211-04 (Other: Arizona Cancer Center - Tucson); UAZ10-16-01 (Other: DCP); N01CN35158 (NIH); P30CA023074 (NIH); NCT01528527 (obsolete NCT alias)
Record Dates: First submitted 2011-09-09; First posted 2011-09-14 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2017-12

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (metformin hydrochloride) (Experimental): Patients receive extended-release metformin hydrochloride PO QD for 4-12 weeks.
  Interventions: Drug: metformin hydrochloride; Other: laboratory biomarker analysis
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD for 4-12 weeks.
  Interventions: Other: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: metformin hydrochloride — Given PO
  Other Names: Glucophage
  Arms: Arm I (metformin hydrochloride)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well metformin hydrochloride works compared to placebo in treating patients with prostate cancer undergoing surgery. Metformin hydrochloride may make some enzymes active. These enzymes may block other enzymes needed for cell growth and stop the growth of tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of 4-12 weeks of metformin (metformin hydrochloride) intervention on cell proliferation in the prostatectomy tissue.

SECONDARY OBJECTIVES:

I. To determine the effect of metformin intervention on prostate tissue bioavailability of metformin.

II. To determine the effect of metformin intervention on apoptosis and angiogenesis in the prostatectomy tissue.

III. To determine the effect of metformin intervention on potential molecular targets of metformin including activated protein kinase (AMPK) activation, mammalian target of rapamycin (mTOR) regulation, and cell cycle regulation in the prostatectomy tissue.

IV. To determine the effect of metformin intervention on changes in systemic hormones and growth factors that have been shown to be modulated by metformin in other patient populations including fasting glucose, fasting insulin, insulin-like growth factor axis, testosterone, and sex hormone binding globulin (SHBG).

V. To determine the effect of metformin intervention on changes in prostate-specific antigen (PSA) levels.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive extended-release metformin hydrochloride orally (PO) once daily (QD) for 4-12 weeks.

ARM II: Patients receive placebo PO QD for 4-12 weeks.

Patients in both arms undergo surgery one day after completion of treatment.

After completion of study treatment, patients are followed up within 30 days of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men will be eligible to this study if they are diagnosed with a histologically confirmed organ-confined adenocarcinoma of the prostate (PCa) treatable by prostatectomy and have a current PSA less than 50 ng/ml
* Have not received chemotherapy and/or radiation for any malignancy (excluding non-melanoma skin cancer and cancers confined to organs with removal as only treatment) in the past 5 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 1.5 times institutional upper limits of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 times institutional ULN
* Creatinine within normal institutional limits
* Willing to use adequate contraception (barrier method, abstinence, subject has had a vasectomy or partner is using effective birth control or is postmenopausal) for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Type I or type II diabetic patients on treatment with any drug for diabetes or participants with fasting glucose >= 126 mg/dL
* History of impaired liver or kidney function
* Participants with a current history of high alcohol consumption (> 3 standard drinks/day) or binge drinking (5 or more drinks) in one session of 1-3 hours
* History of lactic acidosis or at increased risk for lactic acidosis such as patients with unstable or acute congestive heart failure who are at risk of hypoperfusion with hypoxemia
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical composition to metformin
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of acute or chronic metabolic acidosis
* Concurrent use of cationic drugs (e.g., amiloride, digoxin, morphine, procainamide, quinidine, quinine, ranitidine, triamterene, trimethoprim, or vancomycin)
* Concurrent use of non-study metformin or other biguanides

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krouse, Principal Investigator — Arizona Cancer Center - Tucson
Locations (3):
- United States (3):
  - Arizona Cancer Center - Tucson, Tucson, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - University of Southern California/Norris Cancer Center, Los Angeles, California

REFERENCES:
- [Derived] Roy S, Malone S, Grimes S, Morgan SC. Impact of Concomitant Medications on Biochemical Outcome in Localised Prostate Cancer Treated with Radiotherapy and Androgen Deprivation Therapy. Clin Oncol (R Coll Radiol). 2021 Mar;33(3):181-190. doi: 10.1016/j.clon.2020.09.005. Epub 2020 Sep 29. PMID 32994091
- [Derived] Nguyen MM, Martinez JA, Hsu CH, Sokoloff M, Krouse RS, Gibson BA, Nagle RB, Parnes HL, Cordova C, Chow HS. Bioactivity and prostate tissue distribution of metformin in a preprostatectomy prostate cancer cohort. Eur J Cancer Prev. 2018 Nov;27(6):557-562. doi: 10.1097/CEJ.0000000000000394. PMID 28692586

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Metformin Hydrochloride): Patients receive extended-release metformin hydrochloride PO QD (one 500 mg metformin tablet daily for the first week, followed by two 500 mg metformin tablets daily for the second week, and then three 500 mg tablets daily until the day before surgery) for 4-12 weeks.
- Arm II (Placebo): Patients receive placebo PO QD (one placebo tablet daily for the first week, followed by two placebo tablets daily for the second week, and then three placebo tablets daily until the day before surgery) for 4-12 weeks.
Period: Overall Study
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Metformin Hydrochloride): Patients receive extended-release metformin hydrochloride PO QD (one 500 mg metformin tablet daily for the first week, followed by two 500 mg metformin tablets daily for the second week, and then three 500 mg metformin tablets until the day before surgery) for 4-12 weeks.
- Arm II (Placebo): Patients receive placebo PO QD (one placebo tablet daily for the first week, followed by two placebo tablets daily for the second week, and then three placebo tablets until the day before surgery) for 4-12 weeks.
- Total: Total of all reporting groups
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10) | 61 (6) | 63 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cell Proliferation in the Prostatectomy Tissue as Assessed by Ki67 Expression Using Immunohistochemistry (IHC)
Description: Data between the two study groups will be compared using a two-group t-test at a two-sided 0.05 level of significance. If the data are not normally distributed, a non-parametric rank-sum test will be utilized.
Time Frame: 12 weeks
Population: Participants with tissue sections available from prostatectomy
Measure: Median (Inter-Quartile Range); unit: % positively stained nuclei
Groups:
- Arm I (Metformin Hydrochloride): Patients receive extended-release metformin hydrochloride PO QD (one 500 mg metformin tablet daily for the first week, followed by two 500 mg metformin tablets daily for the second week, and then three 500 mg metformin tablets daily until the day before surgery) for 4-12 weeks.
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 8 | 9
% positively stained nuclei | 6.5 [3.33 to 9.33] | 3.67 [2 to 6]
Statistical Analysis 1: Comparison: Arm I (Metformin Hydrochloride) vs Arm II (Placebo); Test type: Other; p = 0.23, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Prostate Tissue Metformin Concentration Levels as Assessed by Liquid Chromatography Tandem Mass Spectrometry
Time Frame: 12 weeks
Population: analysis limited to patients with fresh frozen prostatectomy tissue
Measure: Median (Inter-Quartile Range); unit: ug/g tissue
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 8 | 7
ug/g tissue | 5.71 [2.62 to 16.18] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Arm I (Metformin Hydrochloride) vs Arm II (Placebo); Test type: Other; p < 0.01, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Apoptosis Levels in the Prostatectomy Tissue as Assessed by IHC of Cleaved Caspase 3
Description: Average number of positively stained cells that exhibited nuclear fragmentation from five randomly selected high-power fields (40x) in the tumor region was calculated for each participant
Time Frame: 12 weeks
Population: Participants with tissue sections available from prostatectomy
Measure: Median (Inter-Quartile Range); unit: Number of positive cells
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 8 | 9
Number of positive cells | 0.07 [0.0 to 0.27] | 0.1 [0.0 to 0.27]
Statistical Analysis 1: Comparison: Arm I (Metformin Hydrochloride) vs Arm II (Placebo); Test type: Other; p = 0.77, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Cell Cycle Regulation in the Prostatectomy Tissue as Assessed by IHC of Cyclin D1
Time Frame: 12 weeks
Population: Participants with tissue sections available from prostatectomy
Measure: Median (Inter-Quartile Range); unit: % positive cells
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 8 | 9
% positive cells | 37.5 [20.83 to 59.17] | 13.3 [6.7 to 21.7]
Statistical Analysis 1: Comparison: Arm I (Metformin Hydrochloride) vs Arm II (Placebo); Test type: Other; p = 0.09, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: mTOR Regulation in the Prostatectomy Tissue as Assessed by IHC of Phospho-p70 S6 Kinase (p-p70S6K)
Time Frame: 12 weeks
Population: Participants with tissue sections available from prostatectomy
Measure: Median (Inter-Quartile Range); unit: % positive cells
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 8 | 9
% positive cells | 66.7 [36.67 to 88.33] | 63.3 [39.2 to 80.0]
Statistical Analysis 1: Comparison: Arm I (Metformin Hydrochloride) vs Arm II (Placebo); Test type: Other; p = 0.72, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Angiogenesis in the Prostatectomy Tissue as Assessed by IHC of CD34
Time Frame: 12 weeks
Population: Data were not collected due to budgetary constraints
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: AMPK Activation in the Prostatectomy Tissue as Assessed by IHC of p-AMPK
Time Frame: 12 weeks
Population: Data were not collected due to budgetary constraints
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Cell Cycle Regulation in the Prostatectomy Tissue as Assessed by IHC of Retinoblastoma Protein Phosphorylation (p-pRb)
Time Frame: 12 weeks
Population: Data were not collected due to budgetary constraints
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Changes in Serum PSA
Time Frame: Baseline and 12 weeks
Population: Analysis limited to participants with fasting serum samples
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 8 | 10
% change | -6.53 [-9.45 to 16.76] | 5.98 [-6.91 to 22.98]
Statistical Analysis 1: Comparison: Arm I (Metformin Hydrochloride) vs Arm II (Placebo); Test type: Other; p = 0.63, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Changes in Serum Fasting Insulin
Time Frame: Baseline and 12 weeks
Population: analysis limited to participants with fasting serum samples
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 8 | 10
% change | -11.42 [-33.26 to 16.88] | 5.66 [-10.67 to 22.47]
Statistical Analysis 1: Comparison: Arm I (Metformin Hydrochloride) vs Arm II (Placebo); Test type: Other; p = 0.25, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Changes in Serum IGF-1/IGFBP-3
Time Frame: Baseline and 12 weeks
Population: analysis limited to participants with fasting serum samples
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 8 | 10
% change | 7.07 [-8.51 to 21.77] | -2.24 [-18.2 to 25.71]
Statistical Analysis 1: Comparison: Arm I (Metformin Hydrochloride) vs Arm II (Placebo); Test type: Other; p = 0.46, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Changes in Serum Testosterone
Time Frame: Baseline and 12 weeks
Population: analysis limited to participants with fasting serum samples
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 8 | 10
% change | -16.12 [-20.43 to 3.10] | 2.04 [-16.70 to 28.77]
Statistical Analysis 1: Comparison: Arm I (Metformin Hydrochloride) vs Arm II (Placebo); Test type: Other; p = 0.46, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Changes in Serum SHBG
Time Frame: Baseline and 12 weeks
Population: analysis limited to participants with fasting serum samples
Measure: Median (Inter-Quartile Range); unit: % change
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 8 | 10
% change | 0.48 [-6.64 to 7.19] | -6.49 [-12.43 to 4.33]
Statistical Analysis 1: Comparison: Arm I (Metformin Hydrochloride) vs Arm II (Placebo); Test type: Other; p = 0.36, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Changes in Serum Fasting Glucose
Time Frame: Baseline and 12 weeks
Population: Data were not collected because insulin is a more relevant outcome measure than glucose
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I (Metformin Hydrochloride) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Metformin Hydrochloride) (N=10) | Arm II (Placebo) (N=10)
influenza (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Metformin Hydrochloride) (N=10) | Arm II (Placebo) (N=10)
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Bloating (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Diverticulosis (Gastrointestinal disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0
Chest pain (Cardiac disorders) | 0 | 1
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 0
Increased urinating frequency (Renal and urinary disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Backpain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 1
Sessile polyps in colon and rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pain (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less